CLINICAL TRIAL: NCT01745133
Title: Olux E Foam and Sorilux Foam Combination Therapy for the Maintenance of Treatment Response in Patients With Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leon Kircik, M.D. (Other)
Collaborators: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor-Investigator, Leon Kircik, M.D., Medical Doctor, Derm Research, PLLC
Organization: Derm Research, PLLC (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLX0112
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Psoriasis
Keywords: Olux E foam; Sorilux foam
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene; Clobetasol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- vehicle (Placebo Comparator): clobetasol propionate 0.05% twice a day for two weeks; then vehicle foam twice a day every day for 8 weeks
  Interventions: Drug: vehicle foam
- calcipotriene (Active Comparator): clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day every day for 8 weeks x
  Interventions: Drug: calcipotriene
- calcipotriene + clobetasol propionate (Active Comparator): clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day on weekdays for 8 weeks + clobetasol propionate 0.05% foam twice a day on weekends for 8 weeks
  Interventions: Drug: calcipotriene + clobetasol propionate

INTERVENTIONS:
Drug: vehicle foam — clobetasol propionate 0.05% twice a day for two weeks; then vehicle foam twice a day every day for 8 weeks
  Arms: vehicle
Drug: calcipotriene — clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day every day for 8 weeks
  Other Names: Sorilux foam 0.005% foam
  Arms: calcipotriene
Drug: calcipotriene + clobetasol propionate — clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day on weekdays + clobetasol propionate 0.05% foam twice a day on weekends for 8 weeks
  Other Names: Sorilux foam + Olux E foam
  Arms: calcipotriene + clobetasol propionate

SUMMARY:
The purpose of the study is to investigate if combined use of OLUX-E™ Foam and SORILUX Foam may help "maintain" the therapeutic benefit that is achieved with OLUX-E™ Foam in the treatment of moderate plaque psoriasis.

OLUX-E™ is a medication that contains a corticosteroid delivered in a foam formulation. SORILUX Foam is a foam formulation of calcipotriene. Both medications have been approved by the FDA for treating plaque psoriasis.

DETAILED DESCRIPTION:
This is a single-center, investigator-blind study. Approximately 60 qualified subjects will be enrolled into a 2 week treatment phase where they will receive 2 weeks of treatment with Olux E foam. After 2 weeks treatment, subjects with a PGA of 0 or 1 will be re-randomized into maintenance phase.

Subjects that achieve PGA scores of >2 will be discontinued from the study and will not be randomized. Subjects that achieve PGA scores of 0 or 1 will enter an 8 week maintenance phase where they will be randomized on a 1:1:1 basis to one of the following treatment groups:

* Vehicle foam (BID)
* Sorilux foam (BID)
* Sorilux foam (BID on weekdays) + Olux E foam (BID on weekends)

Subjects will then attend clinic visits at week 6. At week 10 study treatment will be stopped.

The maximum duration of the study is 10 weeks and consists of a Screening/Baseline Visit (Week -0), Re-randomization to maintenance phase visit (Week 2), treatment follow-up visits at Weeks 6, and end of treatment visit at weeks 10.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, 18 years of age or higher. -Female subjects of childbearing potential must have a negative urine pregnancy test within 7 days prior to the first dose of study drug and practice a reliable method of contraception throughout the study [Exception: Female subjects of child bearing potential who are not sexually active are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided they are counseled to remain sexually inactive for the duration of the study and understand the risks involved in getting pregnant during the study.]
* Moderate plaque type psoriasis eligible for topical therapies.
* A Bod Surface Area (BSA) of 3-10%.
* Physician Global Assessment(PGA) score of 3.
* Able to understand study requirements and sign Informed Consent/Health Insurance Portability and Accountability Act forms.

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control, or male subjects planning a pregnancy with their spouse or partner while in the study.
* History of hypocalcaemia or vitamin D toxicity.
* Serious skin condition (other than psoriasis) or uncontrolled medical condition (in the opinion of the investigator).
* Topical steroids, topical immunomodulators, topical vitamin D derivatives, tar, salicylic acid, anthralin or any other topical treatment for psoriasis within 2 weeks of baseline.
* Use of any biologics within 3 months of baseline.
* Use of other systemic psoriasis treatments (ie, oral retinoids, methotrexate, cyclosporine, or other immunomodulators) within 4 weeks of baseline.
* Use of Ultraviolet B light (UVB) or oral psoralen with ultraviolet A (PUVA) within 2 weeks of baseline.
* Skin conditions (e.g. eczema) psoriasis that may interfere with evaluations of psoriasis.
* Known hypersensitivity to Sorilux Foam Ointment or any of its components.
* Known hypersensitivity to Olux E Foam or any of its components.
* Contraindications according to the Sorilux Foam or Olux E Foam package inserts.
* Current drug or alcohol abuse (Investigator opinion).
* Subject unable to commit to all the assessments required by the protocol.
* Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to the Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H Kircik, MD, Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 screen failure
Groups:
- Vehicle 19: clobetasol propionate 0.05% twice a day for two weeks; then vehicle foam twice a day every day for 8 weeks
  vehicle foam: clobetasol propionate 0.05% twice a day for two weeks; then vehicle foam twice a day every day for 8 weeks
- Calcipotriene 20: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day every day for 8 weeks x
  calcipotriene: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day every day for 8 weeks
- Calcipotriene + Clobetasol Propionate 20: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day on weekdays for 8 weeks + clobetasol propionate 0.05% foam twice a day on weekends for 8 weeks
  calcipotriene + clobetasol propionate: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day on weekdays + clobetasol propionate 0.05% foam twice a day on weekends for 8 weeks
Period: Overall Study
Arm/Group | Vehicle 19 | Calcipotriene 20 | Calcipotriene + Clobetasol Propionate 20
Started | 19 | 20 | 19
Completed | 13 | 16 | 15
Not Completed | 6 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle 19 | Calcipotriene 20 | Calcipotriene + Clobetasol Propionate 20 | Total
Number analyzed (Participants) | 19 | 20 | 19 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 19 | 58
  >=65 years | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 10 | 10 | 12 | 32
  Male | 9 | 10 | 07 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 1 | 11
  White | 13 | 16 | 18 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessement
Description: Percentage of participants with clear or almost clear skin on the PGA scale. 0 = clear
  1. = almost clear
  2. = mild
  3. = moderate
  4. = severe
Time Frame: 10 weeks
Measure: Number; unit: percentage of patients
Groups:
- Vehicle 68%: clobetasol propionate 0.05% twice a day for two weeks; then vehicle foam twice a day every day for 8 weeks
  vehicle foam: clobetasol propionate 0.05% twice a day for two weeks; then vehicle foam twice a day every day for 8 weeks
- Calcipotriene 80%: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day every day for 8 weeks x
  calcipotriene: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day every day for 8 weeks
- Calcipotriene + Clobetasol Propionate 79%: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day on weekdays for 8 weeks + clobetasol propionate 0.05% foam twice a day on weekends for 8 weeks
  calcipotriene + clobetasol propionate: clobetasol propionate 0.05% twice a day for two weeks; then calcipotriene 0.005% foam twice a day on weekdays + clobetasol propionate 0.05% foam twice a day on weekends for 8 weeks
Arm/Group | Vehicle 68% | Calcipotriene 80% | Calcipotriene + Clobetasol Propionate 79%
Number analyzed (Participants) | 13 | 16 | 15
percentage of patients | 68 | 80 | 79

ADVERSE EVENTS:
Arm/Group | Vehicle | Calcipotriene 80% | Calcipotriene + Clobetasol Propionate 79%
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 2/20 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=19) | Calcipotriene 80% (N=20) | Calcipotriene + Clobetasol Propionate 79% (N=19)
right hand fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
worsening of burning and itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
small population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes